CLINICAL TRIAL: NCT02595619
Title: Combined Strategy of Renal Replacement Therapy Plus Extracorporeal Carbon Dioxide Removal in Patients With Acute Kidney Injury
Brief Title: Renal Replacement Therapy Plus Extracorporeal Carbon Dioxide Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Vito Fanelli MD, PhD, Assistant Professor, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 0068144
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Acute Kidney Injury
Keywords: AKI; Extracorporeal Carbon Dioxide Removal; Renal Replacement Therapy; Mechanical Ventilation
MeSH Terms: conditions — Acute Kidney Injury | interventions — Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RRT plus ECCO2R (Experimental)
  Interventions: Device: RRT plus ECCO2R

INTERVENTIONS:
Device: RRT plus ECCO2R — Patients with acute kidney injury will be treated with Renal replacement therapy associated to extracorporeal carbon dioxide removal in a single treatment

SUMMARY:
This study aims to assess whether in patients with acute kidney injury (AKI) requiring mechanical ventilation, a strategy that combines renal replacement therapy (RRT) and extracorporeal carbon dioxide removal (ECCO2R) allows reduction of tidal volume and plateau pressure. Systemic Inflammatory Response and Safety Variables will also be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute kidney injury (AKI) requiring renal-replacement therapy and mechanical ventilation of duration ≥ 48 hours

Exclusion Criteria:

* little chance of survival at 24 h (according to clinical judgment), pregnancy, mechanical ventilation with expected duration lower than 48h, age under 18 and over 90

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Achievement of tidal volume reduction to 4 mL/kg while maintaining pH and PaCO2 to ± 20% of baseline values | 72 hours

SECONDARY OUTCOMES:
Evaluation of inflammatory mediators release in plasma samples of patients | 72 hours
  Plasma Concentrations of interleukin 6, interleukin 8, interleukin 1 beta, tumor necrosis factor alpha
Assessment of the changes in pH | 72 hours
Assessment of the changes in PaCO2 | 72 hours
Assessment of the changes in PaO2 | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Italy